CLINICAL TRIAL: NCT00168896
Title: A Randomised Phase II/III Study to Compare the Combination of Carboplatin Plus Irinotecan Vs. the Combination of Carboplatin Plus Etoposide for SCLC in Extensive Disease Stage
Brief Title: A Study for Small Cell Lung Cancer (SCLC) in Extensive Disease Stage
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Pfizer (Industry); Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Haema CBF SCLC UK/AS 01
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-02-14 (Estimated); Status verified 2001-09

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide

INTERVENTIONS:
Drug: Carboplatin plus Irinotecan vs Carboplatin plus Etoposide

SUMMARY:
Comparison of two combination chemotherapies in the treatment of patients with SLCL

DETAILED DESCRIPTION:
Comparison of two combination chemotherapies in the treatment of patients with SLCL

The combination chemotherapies for this study are Carboplatin plus Irinotecan versus Carboplatin plus Etoposide.

ELIGIBILITY:
Inclusion Criteria:

* cytological or histological proven SCLC Stage I or II at 1st diagnosis
* no prior chemotherapy
* measurable tumor disease
* karnofsky performance 70

Exclusion Criteria:

* second malignancy ( except basal cell carcinoma, CA in situ Cervix uteri)
* NYHA III
* chronic diarrhea, obstructive bowel syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286
Dates: Start 2001-10; Study Completion 2006-12

PRIMARY OUTCOMES:
Primary Endpoint:
Documentation of the remission rate ( Phase II)
Determination of progress free time (Phase III)

SECONDARY OUTCOMES:
Secondary Endpoint:
Documentation of progress free time (Phase II)
Documentation of objective remission rate ( Phase III)
Documentation of 1-year survival rate
Documentation of safety of the drug combination

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Principal Investigator — Charité Campus Benjamin Franklin University Clinic
Locations (1):
- Hematology & Oncology Charité CBF Berlin, Germany, Berlin, State of Berlin, Germany